CLINICAL TRIAL: NCT02639702
Title: Switching From Twice-Daily to Once-Daily Clozapine Dosing in Schizophrenia: A Pilot, Double-Blind, Randomized Controlled Trial
Brief Title: Switching From Twice-Daily to Once-Daily Clozapine Dosing in Schizophrenia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Gary Remington, Professor, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 096/2015
Record Dates: First submitted 2015-12-18; First posted 2015-12-24 (Estimated); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Clozapine; Dosing; Once daily; Regimen; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Clozapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Switch group (Experimental): Participants will receive clozapine once daily at evening or bedtime throughout the study period. If a participant takes ≥200 mg of clozapine at a time other than evening/bedtime, half of this dose will be switched to an evening/bedtime regimen on day 0 (baseline), then another half dose will be switched on day 7 (week 1). Participants will receive placebo in place of the clozapine dose that was switched to evening/bedtime.
  Interventions: Drug: Clozapine
- Maintenance group (No Intervention): Participants will continue to take clozapine twice daily throughout the study period.

INTERVENTIONS:
Drug: Clozapine — Switching from twice-daily to once-daily clozapine dosing regimen
  Other Names: Clozaril
  Arms: Switch group

SUMMARY:
Plasma half-life has routinely been used to establish the dosing schedule of antipsychotics; for example, it is recommended that agents with a short plasma half-life be administered multiple times per day. However, to date, several randomized controlled trials (RCTs) have shown no differences in clinical outcomes between once- and twice-daily dosing of various antipsychotics, suggesting that once-daily dosing of antipsychotics is a viable option regardless of plasma half-life. This would apply to clozapine as well; however, there have been no studies comparing once-daily vs. twice-daily dosing regimens of clozapine in terms of efficacy and tolerability. To address this gap in the literature, the investigators shall conduct a pilot, double-blind, RCT to examine efficacy and tolerability following a switch to once-daily dosing regimen of clozapine in patients with schizophrenia receiving clozapine twice a day.

DETAILED DESCRIPTION:
Plasma half-life has routinely been used to establish the dosing schedule of antipsychotics; for example, it is recommended that agents with a short plasma half-life be administered multiple times per day. To date, however, several randomized controlled trials (RCTs) have shown that once-daily dosing of antipsychotics including perphenazine, risperidone, olanzapine, quetiapine, and asenapine is comparable to twice-daily dosing in terms of efficacy and tolerability, suggesting that once-daily dosing of antipsychotics is a viable option regardless of plasma half-life.

This issue applies to clozapine as well, in that it has a relatively short plasma half-life of 12-16 hours; of note, the product monographs recommends that clozapine be administered more than once daily if the dose exceeds 200 mg/day in Canada. Despite this, in clinical practice clozapine is frequently administered once daily because of convenience and side effects such as a daytime sedation or somnolence, In support of this, a cross-sectional survey done at the investigators' own centre has revealed that clozapine was prescribed once daily in 75.1% of 676 patients, even though >200 mg/day was administered in 88.6%. However, there have been no studies comparing once-daily vs. twice-daily dosing regimens of clozapine in terms of efficacy and tolerability. To address this gap in the literature, the investigators shall conduct a pilot, double-blind, RCT to examine efficacy and tolerability following a switch to once-daily dosing regimen of clozapine in patients with schizophrenia receiving clozapine twice a day.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with schizophrenia or schizoaffective disorder based on DSM-IV criteria
* Outpatient status
* Ages 18 years or older
* Has received clozapine twice a day, one of which is in the evening/bedtime, at the same dose and dosing regimen for at least 3 months
* Fluent in English and competent to provide written informed consent

Exclusion Criteria:

* Having significant medical or neurological illnesses
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Brief Psychiatric Rating 18 item Scale (BPRS 18 item scale) | 0 and 12 weeks
  Change in BPRS total scores from baseline to 12 weeks
  Total scores range from 18-126, higher scores represent worse clinical outcomes:
  <31 = Illness not significant >=31 = Mildly ill >41 = Moderately ill >53 = Markedly ill.

SECONDARY OUTCOMES:
Glasgow Antipsychotic Side-effect Scale for Clozapine (GASS-C) | 0 and 12 weeks
  Detect side effects related to Clozapine from baseline to 12 weeks
  Higher Scores indicating worse side-effects:
  0-16 (absent/mild side-effects) 17-32 (moderate side-effects) 33-48 (severe side-effects)
Brief Evaluation of Psychosis Symptom Domains (BE-PSD) | 0 and 12 weeks
  Assess the overall severity of five symptom domains of BE-PSD with a total score in each domain scoring from absent to very severe (i.e. 0-6 with higher scores with worse outcomes)
Personal and Social Performance scale (PSP) | 0 and 12 weeks
  Change in patients social functioning scores from baseline to 12 weeks The PSP is a 100-point single item rating scale from 1-100, subdivided into 10 equal intervals with higher scores indicating better outcomes. The ratings are based on patient's functioning in four main areas: 1) socially useful activities, 2) personal and social relationships, 3) self-care; and 4) disturbing and aggressive behaviours.
Clinical Global Impression - Severity of Illness (CGI-S) | 0 and 12 weeks
  Assess severity of Illness in Schizophrenia CGI scores from baseline to 12 weeks Scores ranging from normal to the most ill (i.e., scores ranging from 1-7 with higher scores with illness worsening)
Brief Neurocognitive Assessment (BNA) | 0 and 12 weeks
  The BNA is a brief neurocognitive assessment that measures global cognitive impairment in patients with schizophrenia from baseline to 12 weeks. Negative Z scores (i.e., -0.5 to -2.0 ) indicate mild to severe cognitive impairment.
Subjective Well-being under Neuroleptics scale - Short form (SWNS) | 0 and 12 weeks
  Self report scale to measure well being. Study assess changes in subjective wellbeing in patients on a neuroleptic from baseline to Week 12. Higher total score indicating better outcomes
Change in the Visual Analogue Scale for Distress Associated with Symptoms (VAS-DAS) scores from baseline to 12 weeks | 0 and 12 weeks
  Assess changes in level of distress associated with symptoms from no distress to worst distress (i.e., 0-100)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Remington, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takeuchi H, Fervaha G, Uchida H, Suzuki T, Bies RR, Gronte D, Remington G. Impact of once- versus twice-daily perphenazine dosing on clinical outcomes: an analysis of the CATIE data. J Clin Psychiatry. 2014 May;75(5):506-11. doi: 10.4088/JCP.13m08695. PMID 24569099
- [Background] Nair NP. Therapeutic equivalence of risperidone given once daily and twice daily in patients with schizophrenia. The Risperidone Study Group. J Clin Psychopharmacol. 1998 Apr;18(2):103-10. doi: 10.1097/00004714-199804000-00002. PMID 9555595
- [Background] Agarwal V, Chadda RK. Once daily risperidone in treatment of schizophrenia. Indian J Psychiatry. 2001 Jan;43(1):32-5. PMID 21407835
- [Background] Takeuchi H, Fervaha G, Lee J, Agid O, Remington G. Effectiveness of different dosing regimens of risperidone and olanzapine in schizophrenia. Eur Neuropsychopharmacol. 2015 Mar;25(3):295-302. doi: 10.1016/j.euroneuro.2014.12.008. Epub 2015 Jan 9. PMID 25649680
- [Background] Chengappa KN, Parepally H, Brar JS, Mullen J, Shilling A, Goldstein JM. A random-assignment, double-blind, clinical trial of once- vs twice-daily administration of quetiapine fumarate in patients with schizophrenia or schizoaffective disorder: a pilot study. Can J Psychiatry. 2003 Apr;48(3):187-94. doi: 10.1177/070674370304800307. PMID 12728743
- [Background] Sun X, Hamer R, McEvoy J. Asenapine once daily versus twice daily: impact on patient acceptance in a randomized, open-label, 14-day clinical trial. J Clin Psychiatry. 2015 Jul;76(7):992-3. doi: 10.4088/JCP.14l09206. No abstract available. PMID 26231009
- [Background] Hiemke C, Baumann P, Bergemann N, Conca A, Dietmaier O, Egberts K, Fric M, Gerlach M, Greiner C, Grunder G, Haen E, Havemann-Reinecke U, Jaquenoud Sirot E, Kirchherr H, Laux G, Lutz UC, Messer T, Muller MJ, Pfuhlmann B, Rambeck B, Riederer P, Schoppek B, Stingl J, Uhr M, Ulrich S, Waschgler R, Zernig G. AGNP Consensus Guidelines for Therapeutic Drug Monitoring in Psychiatry: Update 2011. Pharmacopsychiatry. 2011 Sep;44(6):195-235. doi: 10.1055/s-0031-1286287. Epub 2011 Sep 27. PMID 21969060
- [Background] Takeuchi H, Powell V, Geisler S, DeSanti M, Fervaha G, Agid O, Kane JM, Remington G. Clozapine administration in clinical practice: once-daily versus divided dosing. Acta Psychiatr Scand. 2016 Sep;134(3):234-40. doi: 10.1111/acps.12593. Epub 2016 May 16. PMID 27182769
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.ca/en/research